CLINICAL TRIAL: NCT02754726
Title: A Phase II Pilot Trial of Nivolumab + Albumin-Bound Paclitaxel + Paricalcitol + Cisplatin + Gemcitabine (NAPPCG) In Patients With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Combination Therapy for Patients With Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Translational Genomics Research Institute (Other); Bristol-Myers Squibb (Industry); Lustgarten Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAPPCG-EB 2015-001
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Untreated Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Nivolumab; Albumin-Bound Paclitaxel; paricalcitol; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Other): open label using combination therapy
  Interventions: Drug: Nivolumab; Drug: Albumin-bound paclitaxel; Drug: Paricalcitol; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240mg 240 mg as a 60 minute infusion on days 1, 15, 29 per 42 day cycle
  Other Names: Opdivo
Drug: Albumin-bound paclitaxel — 125 mg/m2 over 30 minutes IV infusion on days 1, 8 and 22, 29 per 42 day cycle
  Other Names: Abraxane
Drug: Paricalcitol — 25 micrograms IV on days 1,4,8,12,15,18,22,26,29,32,36,39 (+/-1 day allowed for dosing per 42 day cycle
  Other Names: Zemplar
Drug: Cisplatin — 25 mg/m2 over 60 minutes IV infusion on days 1, 8 and 22, 29 per 42 day cycle
  Other Names: Platinol
Drug: Gemcitabine — 1000 mg/m2 over 30 minutes IV infusion on days 1, 8 and 22, 29 per 42 day cycle
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to find out if the study drugs nivolumab, albumin- bound paclitaxel, paricalcitol, cisplatin, and gemcitabine given together are safe and effective when combined to treat advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age .
2. Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma.
3. Capable of providing informed consent and complying with Trial procedures.
4. Karnofsky Performance Status (KPS) of ≥ 70%.
5. Life expectancy ≥ 12 weeks.
6. Measurable tumor lesions according to RECIST 1.1 criteria.
7. Women must not be able to become pregnant (e.g. post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating. Both male and female patients of reproductive potential must agree to use a reliable method of birth control during the study.

Exclusion Criteria:

1. Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatments in the adjuvant setting with gemcitabine and/or 5-FU (5-Fluorouracil) or gemcitabine administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
2. Palliative surgery and/or radiation treatment less than 4 weeks prior to initiation of study treatment.
3. Exposure to any investigational agent within 4 weeks prior to initiation of study treatment.
4. Evidence of central nervous system (CNS) metastasis (negative imaging study, if clinically indicated, within 4 weeks of Screening Visit).
5. History of other malignancies (except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix) unless documented free of cancer for ≥5 years.
6. Laboratory values: Screening serum creatinine > upper limit of normal (ULN); total bilirubin > (ULN); alanine aminotransferase (ALT) and Aspartate transaminase (AST) ≥ 2.5 ULN or ≥ 5.0×ULN if liver metastases are present; absolute neutrophil count <1,500/mm3, platelet concentration <100,000/mm3, hematocrit level <27% for females or <30% for males, or coagulation tests (prothrombin time [PT], partial thromboplastin time [PTT], International Normalized Ratio [INR]) >1.5×ULN unless on therapeutic doses of warfarin.
7. Current, serious, clinically significant cardiac arrhythmias as determined by the investigator.
8. History of HIV infection or active or chronic hepatitis B or C.
9. Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals.
10. Major surgery within 4 weeks prior to initiation of study treatment.
11. Any condition that might interfere with the patient's participation in the study or in the evaluation of the study results.
12. Any condition that is unstable and could jeopardize the patient's participation in the study.
13. Patient has a transplanted organ.
14. Patients with a history of autoimmune disease.
15. Prior Programmed cell death protein-1 (PD-1) or Programmed death-ligand-1 (PD-L1) therapy.
16. Patients taking any chemo or immunosuppressive steroids (equivalent to > 20 mg hydrocortisone per day).
17. Patients cannot have > Grade 1 pre-existing peripheral neuropathy (per CTCAE).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Borazanci, MD, Principal Investigator — HonorHealth Research Institute
Locations (1):
- Clinical Trials Nurse Navigator, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 35
Completed | 0
Not Completed | 35
Not completed — Progressive Disease by RECIST | 13
Not completed — Achieved Best Response and converted to maintenance treatment off study | 12
Not completed — Clinical Disease Progression | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Tolerability | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 63.0 [42.0 to 77.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
KARNOFSKY PERFORMANCE STATUS [Count of Participants; unit: Participants] — The Karnofsky Performance Scale Index allows patients to be graded and classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses. The higher Karnofsky score on the scale (0 =unable to care for self, requires equivalent of institutional or hospital care, disease may be progressing; 100=able to carry on normal activity and to work, no special care needed), indicates Normal, no complaints in functional impairment.
  Participants
    100% | 7
    90% | 18
    80% | 7
    70% | 3
Prior Treatment [Number; unit: participants]
  Prior chemotherapy | 4
  Prior radiation | 2
  Prior Surgery | 4
Primary Tumor Location [Number; unit: participants]
  pancreatic head | 13
  pancreatic body | 9
  pancreatic tail | 13
Cancer Antigen (CA) 19-9 at C1/D1 [Count of Participants; unit: Participants]
  Normal (≤ 35) (U/mL) | 5
  Elevated (> 35) (U/mL) | 30
Tumor Markers CA125 or CEA at C1/D1 [Count of Participants; unit: Participants] — Population: CA19-9 Non-secreters
  Participants
    Elevated CA125 and CA19-9 non-secreters: number analyzed (Participants) | 5
    Elevated CA125 and CA19-9 non-secreters | 3
    Elevated CEA and CA19-9 non-secreters: number analyzed (Participants) | 5
    Elevated CEA and CA19-9 non-secreters | 2
Vitamin D, ng/mL [Median (Full Range); unit: ng/mL] | 38.5 [14.2 to 92.6]

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete response (CR) rate as defined by CT scan using RECIST 1.1 criteria - disappearance of all target lesions and no new sites or disease-related symptoms confirmed at least 4 weeks after initial documentation and CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9) down to normal limits; Partial Response (PR), at least a 30% decrease in the sum of the diameters of target lesions; Overall Response (OR) = CR + PR. When a complete response is documented, a Positron emission tomography (PET) scan will be obtained to confirm.
Time Frame: From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 84 months
Population: Not evaluable for overall response as subject did not have post baseline scans (n=3)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 32
Participants
  Overall Response Rate (CR + PR) | 21
  Stable Disease (SD) | 9
  Progressive Disease (PD) | 2

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Patients will be followed throughout their study participation and every 12 weeks following last dose of treatment until reported date of death.
Time Frame: as for outcome 1
Population: adverse events (grade ≥ 3) observed in the study related to study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 35
Participants
  thrombocytopenia | 22
  anemia | 13
  white blood cell decreased | 5
  neutropenia | 4
  peripheral sensory neuropathy | 4
  colitis | 3
  diarrhea | 3
  hypokalemia | 3
  unspecified rash | 3

ADVERSE EVENTS:
Time Frame: 84 months
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 14/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=35)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
colitis (Gastrointestinal disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
diarrhea (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
diverticulitis (Gastrointestinal disorders) | 1 (1)
fever (General disorders) | 1 (1)
joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
leukocytosis (Blood and lymphatic system disorders) | 1 (1)
lung infection (Infections and infestations) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
sepsis (Infections and infestations) | 2 (3)
sinus tachycardia (Cardiac disorders) | 1 (1)
stroke (Nervous system disorders) | 1 (1)
thromboembolic event (Vascular disorders) | 2 (3)
upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=35)
Anemia (Blood and lymphatic system disorders) | 13
Abdominal Pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
alanine aminotransferease increase (Investigations) | 1
neutrophil count decreased (Investigations) | 4
platelet count decreased (Investigations) | 22
white blood cell decreased (Investigations) | 5
diarrhea (Metabolism and nutrition disorders) | 3
hypoalbuminemia (Metabolism and nutrition disorders) | 1
hypokalemia (Metabolism and nutrition disorders) | 3
hypomagnesemia (Metabolism and nutrition disorders) | 1
hyponatremia (Metabolism and nutrition disorders) | 1
hypophosphatemia (Metabolism and nutrition disorders) | 2
vitamin d decreased (Metabolism and nutrition disorders) | 1
peripheral sensory neuropathy (Nervous system disorders) | 4
unspecified rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT02754726/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT02754726/ICF_001.pdf